CLINICAL TRIAL: NCT02987842
Title: Neurofeedback as a Novel Treatment for Mild Cognitive Impairment & Early Alzheimer's
Brief Title: Neurofeedback as a Novel Treatment for Mild Cognitive Impairment & Early Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beersheva Mental Health Center (Other Government)
Responsible Party: Principal Investigator, Doron Todder, Head of anxiety unit, Beersheva Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BeershevaMHC
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
Keywords: Mild cognitive impairment; Alzhiemer's disease; Neurofeedback; EEG
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Patients in the experimental group will receive feedback using the TruScan Neurofeedback system in order to increase the power of EEG in the range of their individual upper alpha (as determined by the peak alpha frequency)
  Interventions: Device: TruScan Neurofeedback
- Sham group (Sham Comparator): Patients in the sham group will receive feedback using the TruScan Neurofeedback system for electrical static activity of a disconnected electrode.
  Interventions: Device: TruScan Neurofeedback

INTERVENTIONS:
Device: TruScan Neurofeedback — Neurofeedback and quantitative EEG system

SUMMARY:
This study protocol proposes an EEG based neurofeedback (EEG-NFB) technique to upregulate the posterior cingulate cortex (PCC) in patients suffering from mild cognitive impairment (MCI) and early Alzheimer's disease (AD).

EEG-NFB has been successfully used as a clinical tool for over 40 years. It is based on electrical activity measured near the surface of the brain using EEG and fed back to the patient within half a second.

MCI is a clinical condition considered as a precursor of AD. NFB appears to be a promising approach to treat MCI, since it has been shown to be able to induce changes in brain plasticity. This research focuses on the PCC, which has been reported to be implicated in MCI, and due to its location (proximity to the surface) accessible by means of EEG- NFB.

A preliminary research in MCI patients, conducted at our lab showed the lower the memory score was at the beginning of the training, the better a subject managed to improve later on. The investigators therefore presume that patients with early Alzheimer's disease, whose cognitive ability is more affected compared to MCI, may benefit from EEG-NFB as well, and maybe to a larger extent compared to MCI.

DETAILED DESCRIPTION:
Cognitive impairment preceding dementia is called mild cognitive impairment (MCI) . Patients with MCI are at high risk for progression to Alzheimer's disease (AD), at a rate of about 12% per year. The amnestic form of MCI is the most common form, and most of the literature on the topic refers to this form of the disorder. Clinical criteria for MCI include:

1. Memory complaint, preferably corroborated by an informant.
2. Objective memory impairment for age and education.
3. Largely intact general cognitive function.
4. Essentially preserved activities of daily living.
5. Not demented

Currently, there is no known cure for MCI or means of stopping or reversing its progression. Patients with Alzheimer's disease were also included in this study , as they are considered by many researchers to be on the same continuum of cognitive decline as patients with MCI which indeed, carry an increased risk for developing Alzheimer's disease.

This study relies the data from a preliminary study conducted in the investigators' lab on patients with MCI, and is meant to further validate our results. In the aforementioned study, participants managed to improve their memory score after 10 training sessions. In addition, a negative correlation between initial memory score and ability to improve was found. It is therefore hypothesized that subjects with AD may benefit as much as subjects with MCI and perhaps even to a larger extent.

Neurofeedback (NFB) is a treatment method based on learning with operant conditioning, in which a feedback (or a reward) is given in proportion with the desired physiological activity in order to improve cognition and/or behavior. This research will focus on using electrical activity measured with EEG as physiological activity to be influenced.

EEG-NFB has been successfully used as a clinical tool for over 40 years treating various disorders from epilepsy, attention deficit hyperactivity disorder (ADHD), stroke to PTSD

Electroencephalography (EEG) equipment is used to measure the electrical activity representing the neuronal activity of different parts of the brain. During the treatment, electrode(s) are placed in predetermined location. Audio and visual rewards are given when the activity is measured to be within the desired frequency range.

Since NFB has been shown to be able to induce changes in the brain plasticity, it appears to be a promising approach to treat MCI. Few studies have shown improvement in cognition of normal elderly with subjective complains of memory decline. To the best of our knowledge, this study is the first to address memory decline in MCI using EEG-based neurofeedback protocol, enhancing the individual upper alpha and peak alpha frequency.

This study will include 30 participants which will be randomly assigned into experimental or sham groups. The former will include training the individual upper alpha, while the latter will include feedback over static electrical activity of a disconnected electrode.

each participant will be trained for a total of 10 sessions over a period of 5 weeks (2 training sessions per week), lasting approx. 1 hour. Cognitive evaluations will take place at baseline, after the training sessions have ended and at 30 days after the last session.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of either mild cognitive impairment or mild Alzheimer's disease
* Age > 50

Exclusion Criteria:

* Active neurological disorder
* Any axis 1 type disorder

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Memory performance | 6 weeks
  improvement in memory performance

SECONDARY OUTCOMES:
General cognitive performance improvement | 6 weeks
  improvement in other cognitive domains
qEEG | 6 weeks
  Improvement in upper alpha to lower alpha power ratio and of peak alpha frequency

CONTACTS AND LOCATIONS:
Overall Officials: Doron Todder, MD/PhD, Principal Investigator — Beersheva Mental Health Center
Locations (1):
- Beer-Sheva Mental Health Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angelakis E, Stathopoulou S, Frymiare JL, Green DL, Lubar JF, Kounios J. EEG neurofeedback: a brief overview and an example of peak alpha frequency training for cognitive enhancement in the elderly. Clin Neuropsychol. 2007 Jan;21(1):110-29. doi: 10.1080/13854040600744839. PMID 17366280
- [Background] Becerra J, Fernandez T, Roca-Stappung M, Diaz-Comas L, Galan L, Bosch J, Espino M, Moreno AJ, Harmony T. Neurofeedback in healthy elderly human subjects with electroencephalographic risk for cognitive disorder. J Alzheimers Dis. 2012;28(2):357-67. doi: 10.3233/JAD-2011-111055. PMID 22002790
- [Background] Jin G, Li K, Hu Y, Qin Y, Wang X, Xiang J, Yang Y, Lu J, Zhong N. Amnestic mild cognitive impairment: functional MR imaging study of response in posterior cingulate cortex and adjacent precuneus during problem-solving tasks. Radiology. 2011 Nov;261(2):525-33. doi: 10.1148/radiol.11102186. Epub 2011 Jul 25. PMID 21788526
- [Background] Panza F, Frisardi V, Capurso C, D'Introno A, Colacicco AM, Chiloiro R, Dellegrazie F, Di Palo A, Capurso A, Solfrizzi V. Effect of donepezil on the continuum of depressive symptoms, mild cognitive impairment, and progression to dementia. J Am Geriatr Soc. 2010 Feb;58(2):389-90. doi: 10.1111/j.1532-5415.2009.02702.x. No abstract available. PMID 20370868
- [Background] Ros T, Munneke MA, Ruge D, Gruzelier JH, Rothwell JC. Endogenous control of waking brain rhythms induces neuroplasticity in humans. Eur J Neurosci. 2010 Feb;31(4):770-8. doi: 10.1111/j.1460-9568.2010.07100.x. PMID 20384819
- [Background] Klimesch W. EEG alpha and theta oscillations reflect cognitive and memory performance: a review and analysis. Brain Res Brain Res Rev. 1999 Apr;29(2-3):169-95. doi: 10.1016/s0165-0173(98)00056-3. PMID 10209231
- [Background] Jelic V, Johansson SE, Almkvist O, Shigeta M, Julin P, Nordberg A, Winblad B, Wahlund LO. Quantitative electroencephalography in mild cognitive impairment: longitudinal changes and possible prediction of Alzheimer's disease. Neurobiol Aging. 2000 Jul-Aug;21(4):533-40. doi: 10.1016/s0197-4580(00)00153-6. PMID 10924766
- [Background] Petersen RC, Caracciolo B, Brayne C, Gauthier S, Jelic V, Fratiglioni L. Mild cognitive impairment: a concept in evolution. J Intern Med. 2014 Mar;275(3):214-28. doi: 10.1111/joim.12190. PMID 24605806
- [Background] Association for Applied Psychophysiology and Biofeedback. Template for developing guidelines for the evaluation of the clinical efficacy of psychophysiological interventions. Appl Psychophysiol Biofeedback. 2002 Dec;27(4):273-81. doi: 10.1023/a:1021061318355. PMID 12557455
- [Background] Zoefel B, Huster RJ, Herrmann CS. Neurofeedback training of the upper alpha frequency band in EEG improves cognitive performance. Neuroimage. 2011 Jan 15;54(2):1427-31. doi: 10.1016/j.neuroimage.2010.08.078. Epub 2010 Sep 17. PMID 20850552